CLINICAL TRIAL: NCT00936234
Title: Functional Improvement of Progenitor Cells and Endothelial Function by Vildagliptin in Diabetes Mellitus (FINNjA-DM).
Acronym: FINNjA-DM
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Florian Seeger, Prof. Dr., Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FINNjA-DM
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: SDF-1 is an Important Cytokine for Neovascularization. Cleavage of SDF-1 is Reduced by DPPIV Inhibitors
Keywords: CAD; diabetes; SDF-1; endothelial function
MeSH Terms: conditions — Diabetes Mellitus | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vildagliptin (Active Comparator): starting with vildagliptin for 30 days followed by placebo for 30 days
  Interventions: Drug: Vildagliptin
- Placebo (Placebo Comparator): starting with placebo for 30 days followed by vildagliptin for 30 days
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin — Vildagliptin, 50 mg twice a days, orally for 30 days followed by placebo
  Other Names: Galvus (R)

SUMMARY:
SDF-1, an important cytokine for neovascularisation is cleaved by (dipeptidyl peptidase IV) DPPIV.

The aim of this study is to assess the effect of the dipeptidyl peptidase IV inhibitor vildagliptin (Galvus®) on endothelial function as well as number and functional activity of progenitor cells in patients with documented diabetes mellitus.

DETAILED DESCRIPTION:
The peptidase CD26 (DPPIV/dipeptidyl peptidase IV) removes dipeptides from the amino terminus of proteins and thereby inactivates these cleaved proteins. It was shown, that CD26 cleaves SDF-1 into a non-mitogenic molecule. Inhibition or deletion of CD26 leads to an increased homing of hematopoietic progenitor cells to the bone marrow after transplantation by increasing the invasion capacity of these cells {Campbell et al. 2008; Christopherson et al. 2004}.

The cytokine SDF-1 is released in response to hypoxia, is crucial for progenitor cell homing and recruitment of cells for neovascularisation. Invasion capacity is closely related to the cytokine SDF-1 and the SDF-1 receptor CXCR4 {Ceradini et al. 2004}. The in vivo neovascularisation capacity of progenitor cells is closely correlated to their functional capacity as SDF-1 induced invasion or colony-forming capacity {Heeschen et al. 2004; Britten et al. 2003; Assmus et al. 2007}.

Therefore, the aim of this study is to assess the effect of the dipeptidyl peptidase IV inhibitor vildagliptin on endothelial function as well as number and functional activity of progenitor cells in patients with documented diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus type 2 under stable medication
* HbA1c between 7% an 10%
* age between 18 and 80 years
* signed informed consent

Exclusion Criteria:

* Atrial fibrillation (plethysmographic recordings can only obtained in sinus-rhythm)
* CAD with reduced left ventricular ejection fraction (LVEF <45%)
* Pregnancy, chronic or acute infection, fever
* Diabetes mellitus type 1
* Newly diagnosed diabetes, uncontrolled diabetes
* Neoplasm
* Known allergy to study drug
* Severe liver/kidney disease
* HIV, Hepatitis
* Participation at other studies within the last 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-09 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | 30 days

SECONDARY OUTCOMES:
Number and Function of Progenitor Cells | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M. Zeiher, MD, Principal Investigator — Cardiology, University of Frankfurt
Locations (1):
- Department of Cardiology, Frankfurt, Germany